CLINICAL TRIAL: NCT01057706
Title: Chiropractic and Exercise Management of Spinal Dysfunction in Seniors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michele Maiers, Faculty, Northwestern Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R18HP15127
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Neck Disability; Back Disability
Keywords: chiropractic; exercise; seniors
MeSH Terms: conditions — Motor Activity | interventions — Manipulation, Chiropractic; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 9 months of chiropractic care and exercise (Experimental): chiropractic, exercise
  Interventions: Other: chiropractic; Behavioral: exercise
- 3 months of chiropractic care and exercise (Active Comparator): chiropractic, exercise
  Interventions: Other: chiropractic; Behavioral: exercise

INTERVENTIONS:
Other: chiropractic — spinal manipulation and mobilization
Behavioral: exercise — strengthening, stretching, balance

SUMMARY:
This study will compare the effectiveness of chiropractic and exercise treatment in the short- and long-term, when managing chronic neck and back disability in seniors over the age of 65 years.

DETAILED DESCRIPTION:
Interventions that temper declining functional status due to aging are critical to the vitality and longevity of the elderly. Conservative, non-drug treatments that address disability and pain may significantly reduce the societal burden associated with spinal dysfunction in this population. Chiropractic and exercise are two such promising therapies, and have yet to be compared in the context of short- versus long-term management.

Unanticipated recruitment challenges and repeated reductions to the award negatively impacted our ability to implement the study as proposed. After careful deliberation among the study's Steering Committee, and approval by the IRB and funding agency, the study has been modified to a 2-treatment comparison (formerly 3 treatments).

As such, the primary aim of this study is to compare the effectiveness of 3 versus 9 months of chiropractic care and exercise in 200 seniors with chronic spinal dysfunction. The primary outcomes are patient-rated neck and back disability.

Additionally, initial inclusion criteria regarding disability ratings have been relaxed to allow more individuals with global spine-related disability to qualify. Specifically, participants now must have:

1. a minimum of 10% disability in both neck and back regions (at least 5/50 on Neck Disability Index (NDI) and Oswestry Disability Index(ODI)) at baseline 1 evaluation, and
2. a combined disability (NDI+ODI) score of at least 25/100 at baseline 1 evaluation.

Secondary aims are to assess between-group differences in patient self-reported pain, general health, improvement, self-efficacy, kinesiophobia, satisfaction, medication use, and objective biomechanical outcomes. Seniors' perceptions and experience with treatment will be assessed through qualitative interviews. Finally, the cost-effectiveness and cost-utility of these interventions will be measured.

Additional secondary aims include assessing within group differences in an additional 18 patients randomized to receive 9 months of exercise only in the earlier phase of this study. Outcomes of these aims include the self-report, biomechanical, and qualitative outcomes listed above (with the exception of cost-effectiveness and cost-utility data).

This project will significantly contribute to the evidence base of conservative, non-drug treatments that address disability and pain in seniors with spinal dysfunction. Identification of effective therapies has tremendous potential to substantially improve the functional status, quality of life, and overall health in the aging population.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* independent ambulation and community dwelling
* stable medication plan
* neck-related disability (minimal score of 10% on Neck Disability Index)
* back-related disability (minimal score of 10% on Oswestry Disability Index)
* minimum combined disability score (above) of 25% at first baseline screening
* at least 12 week duration of neck and back related disability

Exclusion Criteria:

* moderate or severe cognitive impairment
* untreated clinical depression
* surgical spinal fusion or multiple incidents of spinal surgery
* contraindications to spinal manipulation or exercise
* ongoing, non-pharmacological treatment for a spinal condition

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patient-rated neck and back disability | 9 months

SECONDARY OUTCOMES:
Pain | 9 and 18 months
Improvement | 9 and 18 months
General health | 9 and 18 months
Medication use | 9 and 18 months
Satisfaction | 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Maiers, DC, MPH, Principal Investigator — Northwestern Health Sciences University
Locations (1):
- Northwestern Health Sciences University, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Maiers M, Hartvigsen J, Evans R, Westrom K, Wang Q, Schulz C, Leininger B, Bronfort G. Short- or Long-Term Treatment of Spinal Disability in Older Adults With Manipulation and Exercise. Arthritis Care Res (Hoboken). 2019 Nov;71(11):1516-1524. doi: 10.1002/acr.23798. PMID 30354023
- [Derived] Vihstadt C, Maiers M, Westrom K, Bronfort G, Evans R, Hartvigsen J, Schulz C. Short term treatment versus long term management of neck and back disability in older adults utilizing spinal manipulative therapy and supervised exercise: a parallel-group randomized clinical trial evaluating relative effectiveness and harms. Chiropr Man Therap. 2014 Jul 23;22:26. doi: 10.1186/s12998-014-0026-7. eCollection 2014. PMID 25478141